CLINICAL TRIAL: NCT03660397
Title: Efficacy and Safety of Adrenal Artery Ablation（AAA）in the Treatment of Uncontrolled Hypertension: A Randomized, Parallel, Active-controlled Clinical Trial
Brief Title: Adrenal Artery Ablation for Uncontrolled Hypertension
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Zhiming Zhu, Director of the Department of Hypertension & Endocrinology, Daping Hospital, Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAA-UHT
Record Dates: First submitted 2018-06-07; First posted 2018-09-06 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Uncontrolled Hypertension
Keywords: Uncontrolled Hypertension; Resistant hypertension; Aldosterone; Ablation; Adrenal Gland

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Selective endovascular chemical ablation of adrenal gland after adrenal angiography.
  Interventions: Procedure: Selective endovascular chemical ablation of adrenal gland; Drug: Traditional triple antihypertensive treatment
- Control (Active Comparator): No intervention, but treated with standard antihypertensive drugs
  Interventions: Drug: Traditional triple antihypertensive treatment

INTERVENTIONS:
Procedure: Selective endovascular chemical ablation of adrenal gland — Intervention with selective endovascular chemical ablation of adrenal gland is performed after adrenal angiography in the group.
  Arms: Intervention
Drug: Traditional triple antihypertensive treatment — irbesartanhydrochlorothiazide 162.5 mg/d, amlodipine 5 mg/d

SUMMARY:
The activation of the renin-angiotensin-aldosterone system (RAAS) plays a key role in uncontrolled hypertension or resistant hypertension. Surgery and and medicine are the main treatment for primary aldosteronism(PA) by the current guidelines. However, only a small part of patients with PA meet the surgical criteria, and most of patients with uncontrolled hypertension and activation of RAAS have to take spironolactone or other antihypertensive drugs for long time. On the other side, long-term inhibition of aldosterone receptor may cause hyperkalemia, male breast hyperplasia and other adverse reactions. Moreover, hyperaldosterone is still not corrected by spironolactone, which causes extensive cerebrovascular damages even though blood pressure and blood potassium had been normalized.

With the development of adrenal vein sampling and adrenal ablation, selective arterial ablation of adrenal gland(AAA) was observed with significant decrease of blood aldosterone and blood pressure in patients with PA, which made it promising that uncontrolled hypertension could be relieved by selective AAA.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged between 30-60 years old.
* Patients with poorly controlled hypertension (office blood pressure ≥130/80 mmHg) with rational lifestyle change and triple antihypertensive drugs (irbesartanhydrochlorothiazide 162.5 mg/d, amlodipine 5 mg/d) for at least 2 weeks
* Positional blood aldosterone ≥100pg/ml.
* Informed consent signed and agreed to participate in this trial.

Exclusion Criteria:

* Hyperkalemia or hypokalemia.
* Secondary hypertension.
* History of depression, schizophrenia or vascular dementia.
* Renal failure or the following history of nephropathy: serum creatinine 1.5 times higher than the upper limit; dialysis history; or nephrotic syndrome.
* Adrenergic insufficiency.
* Heart failure with NYHA grade Ⅱ-Ⅳ grade or unstable angina, severe cardiovascular and cerebrovascular stenosis, myocardial infarction, intracranial aneurysm, stroke and other acute cardiovascular events.
* Acute infections, tumors and severe arrhythmias, psychiatric disorders,
* drugs or alcohol addicts.
* Liver dysfunction or the following history of liver disease: AST or ALT 3 times higher than the upper limit, liver cirrhosis, history of hepatic encephalopathy, esophageal variceal history or portal shunt history.
* Fertile woman without contraceptives.
* Coagulation dysfunction.
* Pregnant women or lactating women.
* Participated in other clinical trials or admitted with other research drugs within 3 months prior to the trial.
* Any surgical or medical condition which can significantly alter the absorption, distribution, metabolism, or excretion of any study drug.
* Allergy or any contraindications for the study drugs, contrast agents and alcohol.
* Refused to sign informed consent

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-07-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Change of 24-h average systolic blood pressure measured at baseline and the end of the trial | 24 weeks
  Difference in the change of 24-h average systolic blood pressure between the intervention and control group is to be analysed.

SECONDARY OUTCOMES:
Change of 24-h average systolic blood pressure compared with the baseline | 24 weeks
  Change of 24-h average systolic blood pressure compared with the baseline at the end of the study (24 weeks) in the intervention group.
Change of anti-hypertensive regimen measured at baseline and the end of the trial | 24 weeks
  Difference in the change of anti-hypertensive regimen between the intervention and control group is to be analysed.
Change of 24-h average diastolic blood pressure, daytime mean systolic blood pressure, daytime mean diastolic blood pressure, and nighttime average systolic and diastolic blood pressure measured at baseline and the end of the trial | 24 weeks
  Difference in the change of 24-h average diastolic blood pressure, daytime mean systolic blood pressure, daytime mean diastolic blood pressure, and nighttime average systolic and diastolic blood pressure between the intervention and control group is to be analysed.
Change of home systolic and diastolic pressure measured at baseline and the end of the trial | 24 weeks
  Difference in the change of home systolic and diastolic pressure between the intervention and control group is to be analysed.
Change of office systolic and diastolic pressure measured at baseline and the end of the trial | 24 weeks
  Difference in the change of office systolic and diastolic pressure between the intervention and control group is to be analysed.
Change of blood electrolytes measured at baseline and the end of the trial | 24 weeks
  Difference in the change of blood electrolytes between the intervention and control group is to be analysed.
Change of plasma and urine adrenal hormones measured at baseline and the end of the trial | 24 weeks
  Difference in the change of plasma and urine adrenal hormones between the intervention and control group is to be analysed.
Change of plasma renin measured at baseline and the end of the trial | 24 weeks
  Difference in the change of plasma renin between the intervention and control group is to be analysed.
Change of liver enzymes measured at baseline and the end of the trial | 24 weeks
  Difference in the change of liver enzymes (ALT, AST in IU/L) between the intervention and control group is to be analysed.
Change of kidney function measured at baseline and the end of the trial | 24 weeks
  Difference in the change of serum creatinine in umol/L between the intervention and control group is to be analysed.
Change of fasting blood glucose measured at baseline and the end of the trial | 24 weeks
  Difference in the change of fasting blood glucose in mmol/L between the intervention and control group is to be analysed.
Change of lipids profiles measured at baseline and the end of the trial | 24 weeks
  Difference in the change of lipids profiles (TC, HDL-C, LDL-C, TG) in mmol/L between the intervention and control group is to be analysed.

OTHER OUTCOMES:
Change of sex hormones measured at baseline and the end of the trial | 24 weeks
  Difference in the change of 17-OH, DHEAS, testosterone and estrogen levels between the intervention and control group is to be analysed.
Change of 24-h urine microalbumin measured at baseline and the end of the trial | 24 weeks
  Difference in the change of 24-h urine microalbumin, microalbumin/creatinine ratio between the intervention and control group is to be analysed.
Change of echocardiography measured at baseline and the end of the trial | 24 weeks
  Difference in the change of cardiac parameters assessed by echocardiography (IVSd、IVSs、LVPWd, LVPWs, LVEDD, in millimetre(mm), and LVEF(%), LVM in gram) between the intervention and control group is to be analysed.
Change of carotid intima-media thickness assessed by carotid ultrasound at baseline and the end of the trial | 24 weeks
  Difference in the change of carotid intima-media thickness(CIMT) assessed by carotid ultrasound between the intervention and control group is to be analysed.

CONTACTS AND LOCATIONS:
Locations (1):
- The third hospital affiliated to the Third Military Medical University, Chongqing, Chongqing Municipality, China